CLINICAL TRIAL: NCT00485771
Title: Olanzapine/Fluoxetine Combination Versus Lamotrigine in the Treatment of Bipolar I Depression
Brief Title: Olanzapine/Fluoxetine Combination Versus Comparator in the Treatment of Bipolar I Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7980; H6P-US-HDAQ
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Fluoxetine; Lamotrigine

INTERVENTIONS:
Drug: Olanzapine
Drug: Fluoxetine
Drug: Lamotrigine

SUMMARY:
The purpose of this study is to assess olanzapine/fluoxetine combination and lamotrigine comparative efficacy, safety and tolerability in acute and longer term treatment of bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 to 60 years of ages, inpatients or outpatients. Inpatients are qualified only if they are hospitalized for current episode of bipolar depression and should be able to leave hospital when clinical criteria are no longer met for acute inpatient hospitalization
* Patients must fulfill the criteria for bipolar I depression (bipolar I disorder, current episode major depressive) as defined in DSM-IV-TR based on clinical examination and psychiatric assessment
* Patients must have experienced, in the opinion of the investigator, at least one previous manic or mixed episode as defined in DSM-IV-TR, of sufficient severity to require treatment with a mood stabilizer or an antipsychotic as reported by the patient or the caregiver
* Each patient must have a level of understanding sufficient to perform all tests and examinations required by the protocol
* Female patients must test negative for pregnancy and must be using a medically accepted means of contraception

Exclusion Criteria:

* Current diagnosis of any of the following according to DSM-IV-TR criteria: Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder, Delusional Disorder, Delirium of any type, Dementia of any type, Amnestic Disorder, any Substance-Induced Disorder, or any Psychotic Disorder due to a General Medical Condition, unless there is substantive reason to believe patient was previously misdiagnosed.
* Treatment with clozapine within 3 months (90 days) prior to visit 1
* Treatment with electroconvulsive therapy (ECT) within 3 months (90 days) prior to visit 2
* Patients with seizure disorders are excluded (except patients with a previous history of seizures due to alcohol withdrawal, which have resolved).
* Participation in a clinical trial of another drug including olanzapine, fluoxetine or lamotrigine within 30 days prior to study entry (visit 1)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 403 (Actual)
Dates: Start 2003-11; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of olanzapine/fluoxetine combination compared with lamotrigine in the treatment of patients with bipolar I depression during the first 7 weeks of therapy.

SECONDARY OUTCOMES:
Assess the efficacy of olanzapine/fluoxetine combination compared with lamotrigine on depressive symptoms
Assess the onset of action of olanzapine/fluoxetine combination compared with lamotrigine as measured by time to achieve an initial response
Assess the study-defined response and remission rates including time to achieve a full response and time to achieve remission as well as time to sustained response and sustained remission
Assess the time to and rate of relapse to depressive episode following remission for olanzapine/fluoxetine combination compared with lamotrigine
Assess the time to and rate of relapse to mania with olanzapine/fluoxetine combination compared with lamotrigine
Assess efficacy of treatment in improving symptomatology
Evaluate the level of health resource utilization and resource utilization costs associated with olanzapine/fluoxetine combination compared with lamotrigine during the study treatment period
Assess the efficacy of olanzapine/fluoxetine combination compared with lamotrigine for suicide ideation
Assess the total time of hospitalization of patients on olanzapine/fluoxetine combination compared with lamotrigine during the study treatment period
Assess the safety and tolerability of olanzapine/fluoxetine combination compared with lamotrigine during 6 months of therapy
The sensitivity and positive predictive value of the MDQ will be determined in this study, using the SCID as a standard
To explore possible correlation between changes in eating behavior and changes in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana, United States

REFERENCES:
- [Derived] Houston J, Dharia S, Bishop JR, Ellingrod VL, Fijal B, Jacobson JG, Hoffmann VP. Association of DRD2 and ANKK1 polymorphisms with prolactin increase in olanzapine-treated women. Psychiatry Res. 2011 May 15;187(1-2):74-9. doi: 10.1016/j.psychres.2010.10.020. Epub 2010 Nov 20. PMID 21095016
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com